CLINICAL TRIAL: NCT05794971
Title: Regorafenib Combined With Irinotecan Drug-Eluting Beads as Third-line Treatment for Colorectal Cancer Liver Metastases: a Multicentre, Randomised Phase 3 Trial (RIDER)
Brief Title: Regorafenib Combined With Irinotecan Drug-Eluting Beads for Colorectal Cancer Liver Metastases
Acronym: RIDER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director of Medical Oncology, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-IC-01
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer Liver Metastases; Regorafenib
MeSH Terms: interventions — regorafenib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan Drug-Eluting Beads combined with regorafenib (Experimental)
  Interventions: Drug: Regorafenib and DIBIRI
- regorafenib (Active Comparator)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib and DIBIRI — Drug: Regorafenib Regorafenib will be given 3 weeks on/1 week off (initial dose: 80 mg od po.)
  Drug: Irinotecan it will be mixed in eluting-beads and injected in the tumor.
  Procedure: TACE Transcatheter arterial chemoembolization（TACE）is a minimally invasive procedure performed to decrease the tumor's blood supply.
  Device: drug eluting-bead The eluting-bead,loaded with irinotecan (DEBIRI) to treat patients with hepatic metastases from colorectal cancer.
  Other Names: Drug: Irinotecan; Procedure: TACE; Device: drug eluting-bead
  Arms: Irinotecan Drug-Eluting Beads combined with regorafenib
Drug: Regorafenib — Drug: Regorafenib Regorafenib will be given 3 weeks on/1 week off (initial dose: 80 mg od po.)
  Arms: regorafenib

SUMMARY:
This study is a multicentre, prospective, randomised trial, aims to evaluate the efficacy and safety of Irinotecan Drug-Eluting Beads combined with regorafenib as the third-line treatment for a patient with colorectal cancer liver metastases. The study is planned to enrolled 126 patients failing first- and second-line standard chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, of any race or sex, who have histologic or radiologic proof of colorectal cancer to the liver, who are able to give informed consent, will be eligible.
* Patients failing first- and second-line standard systemic chemotherapy.
* Patients with at least one measurable liver metastases, with size > 1cm response evaluation criteria in solid tumors (RECIST)
* Patients with liver dominant disease defined as ≥80% tumor body burden confined to the liver
* Less than 60% liver tumor replacement
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of < 2
* Child-pugh's grade A or B
* Life expectancy of > 3 months
* Non-pregnant with an acceptable contraception in premenopausal women.
* Hematologic function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, white cell count (WBC) ≥ 3.0 x 109/L, platelets ≥75 x109/L, international normalized ratio (INR) ≤1.3.
* Adequate hepatic and renal function: Alanine aminotransferase (ALT) or aspartate aminotransferase ≤2.5×above upper normal range, total bilirubin≤1.5×above upper normal range, Serum creatinine≤1.5×above upper normal range
* Women of child bearing potential and fertile men are required to use effective contraception negative serum beta human chorionic gonadotropin (βHCG)
* Signed, written informed consent

Exclusion Criteria:

* Prior treatment with TACE, regorafenib or fruquintinib
* Patients with brain metastases
* With serious heart, kidney, bone marrow, or lung, central nervous system diseases.
* Patients suffered with other cancer.
* patients who were seriously ill and had history of chronic disease such as tuberculosis (TB) and human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS) were excluded from the study.
* known or suspected history of allergy to any of the related drugs used in the study
* Women who are pregnant or breast feeding
* Patients with serious somatic or psychiatric illness regarded as contraindications or in need of treatment that would interfere with study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 24 months
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  The PFS is defined as the time from the start of treatment to the date of first documented PD or death as a result of any cause, whichever occurred first. When a patient was alive and without progression, PFS was censored at the date of the last disease assessment.
Objective Response Rate (ORR) | 24 months
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)
Disease Control Rate (DCR) | 24 months
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD); CR, PR, or SD had to be maintained for at least 28 days from the first demonstration of that rating)
Duration of response (DOR) | 24 months
  It was defined as the time from the first judgment of complete remission (CR) or partial remission (PR) to the discovery of disease progression (PD) after treatment
Adverse enents | 24 months
  Safety variables will be summarized using descriptive statistics based on adverse events collection

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhang, M.D, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Bo Zhang, Guangdong, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No